CLINICAL TRIAL: NCT02354391
Title: Ingenol Mebutate (Picato®) With Methyl Aminolevulinate Photodynamic Therapy for the Treatment of Actinic Keratosis.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Pacific Dermaesthetics (Other)
Collaborators: LEO Pharma (Industry)
Responsible Party: Principal Investigator, Jason K Rivers, MD, FRCPC, FAAD, Principal Investigator, Pacific Dermaesthetics
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1969699
Record Dates: First submitted 2015-01-20; First posted 2015-02-03 (Estimated); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Actinic Keratosis
MeSH Terms: conditions — Keratosis, Actinic | interventions — 3-ingenyl angelate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ingenol mebutate and MAL PDT (Experimental): Participants will recieve Ingenol mebutate 0.015% topical gel treatment applied day 2,3 and 4 to quadrant 1. Patients will recieve ingenol mebutate 0.015% applied on day 1 followed by methyl aminolevulate and photodyamnic therapy on day 5 to quadrant 2. Particpants will recieve methyl aminolevulate and photodynamic therapy on day 5 to quadrant 3, and quadrant 4 will act as the control, with no treatment.
  Interventions: Drug: Ingenol mebutate Picato® and MAL PDT day 1, day 5; Drug: Ingenol mebutate Picato® day 2, 3, 4; Procedure: MAL PDT day 5

INTERVENTIONS:
Drug: Ingenol mebutate Picato® and MAL PDT day 1, day 5 — Treatment of ingenol mebutate, Picato® 0.015% topical gel applied on day 1 followed by MAL PDT on day 5
  Other Names: Picato® 0.015% and MAL PDT
Drug: Ingenol mebutate Picato® day 2, 3, 4 — Full treatment course with Ingenol mebutate (Picato®) 0.015% topical gel, apply day 2,3 and 4
  Other Names: Picato® 0.015%
Procedure: MAL PDT day 5 — Methyl aminolevulate combined with Photodynamic therapy at day 5
  Other Names: MAL PDT

SUMMARY:
The objective of this study is to determine the efficacy, safety, and patient satisfaction of pretreatment with Picato® gel 4 days prior to methyl aminolevulinate photodynamic therapy (MAL PDT). Patients diagnosed with actinic keratosis who are eligible to receive topical treatment with ingenol mebutate (Picato®) and photodynamic therapy will act both as the test group and the control group. Each patient will have four distinct treatment areas of 25cm2 on the scalp, and/or scalp and face. Three of the treatment areas will receive Picato® 0.015% gel, MAL PDT, or Picato® 0.015% and MAL PDT combined. One area will serve as a control and will receive none of the treatments.

DETAILED DESCRIPTION:
Study Objective The objective of this study is to determine the efficacy, safety and patient satisfaction of pretreatment with Picato® gel 4 days prior to methyl aminolevulinate photodynamic therapy (MAL PDT). This test area will be compared to Picato® treatment alone or MAL PDT alone treatment areas as well as a control field (no treatment).

Rationale This study focuses on the topical treatment of actinic keratosis. Patients diagnosed with actinic keratosis who are eligible to receive topical treatment with ingenol mebutate (Picato®) and photodynamic therapy will act both as the test group and the control group. Patients will be followed through appointments with the study nurse and dermatologist.

Patient treatment eligibility and regimen for prescribed medication are at Dr. Rivers (and patient's) discretion. Patients will be followed in the study for the duration of one complete treatment plus 2 months.

Study duration:

The inclusion period is 6 months, depending on the speed of patient recruitment. The study duration for each individual patient will end eight weeks after treatment completion.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 40 yrs
2. Patients eligible to receive topical treatment with ingenol mebutate gel and photodynamic therapy for treatment of actinic keratosis at the discretion of the dermatologist.
3. Fitzpatrick Skin Type I & II.
4. Patient must give informed consent.

Exclusion Criteria:

1. Diagnosis of Basal Cell Carcinoma(BCC), Squamous Cell Carcinoma(SCC) or melanoma in the treatment area.
2. Currently experiencing adverse reactions and/or Local Skin Reactions from previous Actinic Keratosis(AK) treatment in the treatment field.
3. Females who are pregnant, nursing or planning a pregnancy during their participation in the study.
4. Female subjects of childbearing potential (including subjects using surgical sterilization, ie, bilateral tubal ligation or implanted device methods of contraception) with a positive urine pregnancy test at Day 1 prior to study treatment; a female is considered NOT to be of childbearing potential if she is post-menopausal with at least 12 consecutive months of amenorrhea, has undergone bilateral oophorectomy, or has no uterus.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-01; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Complete clearance of lesions | 60 days
  The proportion of patients with complete clearance of actinic keratoses in the treatment area compared to baseline.

SECONDARY OUTCOMES:
Localized skin response to Erythema is measured using a 4 point scale, 0 (no erythema) to 3 (severe erythema) | Day 5, 8 and 15
  Assessment of erythema as part of an evaluation of tolerance of 3 treatments: Ingenol mebutate 0.015% topical gel, MAL PDT, and Ingenol mebutate 0.05% topical gel combined with MAL PDT. This will be done by visual assessment by the Investigator using a 4 point scale. The scale is 0=none present, 1=mild , 2=moderate, and 3=severe.
Count of actinic kertosis lesions | 60 days (day 15, 30 and 60)
  The percent change in actinic keratosis count as compared to the baseline lesion count.
Localized skin response to Flaking/Scaling is measured using a 4 point scale, 0 (no flaking/scaling) to 3 (severe flaking/scaling) | Day 5, 8 and 15
  Assessment of Flaking/Scaling as part of an evaluation of tolerance of 3 treatments: Ingenol mebutate 0.015% topical gel, MAL PDT, and Ingenol mebutate 0.05% topical gel combined with MAL PDT. This will be done by visual assessment by the Investigator using a 4 point scale. The scale is 0=none present, 1=mild , 2=moderate, and 3=severe.
Localized skin response to Pustulation is measured using a 4 point scale, 0 (no pustulation) to 3 (severe pustulation) | Day 5, 8 and 15
  Assessment of Pustulation as part of an evaluation of tolerance of 3 treatments: Ingenol mebutate 0.015% topical gel, MAL PDT, and Ingenol mebutate 0.05% topical gel combined with MAL PDT. This will be done by visual assessment by the Investigator using a 4 point scale. The scale is 0=none present, 1=mild , 2=moderate, and 3=severe.
Localized skin response to Vesiculation is measured using a 4 point scale, 0 (no vesiculation) to 3 (severe vesiculation) | Day 5, 8 and 15
  Assessment of Vesiculation as part of an evaluation of tolerance of 3 treatments: Ingenol mebutate 0.015% topical gel, MAL PDT, and Ingenol mebutate 0.05% topical gel combined with MAL PDT. This will be done by visual assessment by the Investigator using a 4 point scale. The scale is 0=none present, 1=mild , 2=moderate, and 3=severe.
Localized skin response to Pain is measured using a 4 point scale, 0 (no pain) to 3 (severe pain) | Day 5, 8 and 15
  Assessment of Pain as part of an evaluation of tolerance of 3 treatments: Ingenol mebutate 0.015% topical gel, MAL PDT, and Ingenol mebutate 0.05% topical gel combined with MAL PDT. This will be done by visual assessment by the Investigator using a 4 point scale. The scale is 0=none present, 1=mild , 2=moderate, and 3=severe.
Localized skin response to Crusting is measured using a 4 point scale, 0 (no crusting) to 3 (severe crusting) | Day 5, 8 and 15
  Assessment of Crusting as part of an evaluation of tolerance of 3 treatments: Ingenol mebutate 0.015% topical gel, MAL PDT, and Ingenol mebutate 0.05% topical gel combined with MAL PDT. This will be done by visual assessment by the Investigator using a 4 point scale. The scale is 0=none present, 1=mild , 2=moderate, and 3=severe.
Localized skin response to Swelling is measured using a 4 point scale, 0 (no swelling) to 3 (severe swelling) | Day 5, 8 and 15
  Assessment of Swelling as part of an evaluation of tolerance of 3 treatments: Ingenol mebutate 0.015% topical gel, MAL PDT, and Ingenol mebutate 0.05% topical gel combined with MAL PDT. This will be done by visual assessment by the Investigator using a 4 point scale. The scale is 0=none present, 1=mild , 2=moderate, and 3=severe.
Localized skin response to Erosion/Ulceration is measured using a 4 point scale, 0 (no erosion/ulceration) to 3 (severe erosion/ulceration) | Day 5, 8 and 15
  Assessment of Erosion/Ulceration as part of an evaluation of tolerance of 3 treatments: Ingenol mebutate 0.015% topical gel, MAL PDT, and Ingenol mebutate 0.05% topical gel combined with MAL PDT. This will be done by visual assessment by the Investigator using a 4 point scale. The scale is 0=none present, 1=mild , 2=moderate, and 3=severe.
VAS questionnaire - How much pain was associated with the use of Picato® for 3 days? | Day 5
  Participants will be presented with a questionnaire at day 5 asking: How much pain was associated with the use of Picato® for 3 days? Participants will answer using the 0-10 VAS Numeric Pain Distress Scale (0 = no pain, 5 = moderate pain, 10 = unbearable pain).
VAS questionnaire - How much pain was associated with the use of Picato® followed by PDT? | Day 5
  Participants will be presented with a questionnaire at day 5 asking: How much pain was associated with the use of Picato® followed by PDT? Participants will answer using the 0-10 VAS Numeric Pain Distress Scale (0 = no pain, 5 = moderate pain, 10 = unbearable pain).
VAS questionnaire - How much pain did you experience in the PDT treatment area? | Day 5
  Participants will be presented with a questionnaire at day 5 asking:How much pain did you experience in the PDT treatment area? Participants will answer using the 0-10 VAS Numeric Pain Distress Scale (0 = no pain, 5 = moderate pain, 10 = unbearable pain).
Patient Assessment Questionnaire - Patient evaluation of the following treatments: Ingenol mebutate 0.015% topical gel, MAL PDT, and Ingenol mebutate 0.05% topical gel combined with MAL PDT. | Day 15
  Patients will be asked to evaluate each of the treatments they have received (Ingenol mebutate 0.015% topical gel, MAL PDT, and Ingenol mebutate 0.05% topical gel combined with MAL PDT). They will be presented with a questionnaire at Day 15 asking the following questions:
  1. Would you used this treatment again? (Yes, No)
  2. Talking all things into account, how satisfied or dissatisfied with the outcome of using this medication? (Very dissatisfied, Dissatisfied, Somewhat Satisfied, Satisfied, Extremely Satisfied)
  3. How does this treatment compare to the other treatments? (Worse, Slightly Worse, No Change, Slightly Better, Much Better)